CLINICAL TRIAL: NCT06191471
Title: Hepatitis A Virus Induced Acute Acalculous Cholecystitis Diagnosed Postoperatively: Case Report
Status: Completed | Type: Observational
Sponsor: University of Balamand (Other)
Responsible Party: Principal Investigator, Omar Tabbikha, Resident doctor, University of Balamand
Other Study IDs: UBalamandAAC
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Acute Acalculous Cholecystitis
Keywords: Acute acalculous cholecystitis
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gallbladder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laparoscopic cholecystectomy for hepatitis A induced acute acalculous cholecystitis — Laparoscopic cholecystectomy for hepatitis A induced acute acalculous cholecystitis

SUMMARY:
41-year-old previously healthy patient presented with right upper quadrant abdominal pain. Pain started two days prior to presentation when an abdominal ultrasound in a peripheral hospital showed a 10 mm gallbladder stone with normal laboratory tests; however, her pain was resolved on analgesics. Now the pain was persistent and associated with vomiting and laboratory tests showed elevated bilirubin. Laparoscopic cholecystectomy with intraoperative cholangiography was done that showed inflamed gallbladder but with no stones and normal cholangiography. Day one post-operation, while the pain resolved, labs showed elevated liver function tests and hepatitis workup showed acute HAV infection attributing her presentation to HAV induced AAC.

DETAILED DESCRIPTION:
Introduction: acute acalculous cholecystitis (AAC) is defined as gallbladder inflammation without the presence of stones. Contrary, hepatitis A virus (HAV) causes acute hepatitis A and can present with different symptoms; however, HAV causing and presenting as AAC is rare.

Case presentation: 41-year-old previously healthy patient presented with right upper quadrant abdominal pain. Pain started two days prior to presentation when an abdominal ultrasound in a peripheral hospital showed a 10 mm gallbladder stone with normal laboratory tests; however, her pain was resolved on analgesics. Now the pain was persistent and associated with vomiting and laboratory tests showed elevated bilirubin. Laparoscopic cholecystectomy with intraoperative cholangiography was done that showed inflamed gallbladder but with no stones and normal cholangiography. Day one post-operation, while the pain resolved, labs showed elevated liver function tests and hepatitis workup showed acute HAV infection attributing her presentation to HAV induced AAC.

Discussion: AAC is usually caused by stasis of the gallbladder due to different causes; however, HAV as the cause of AAC has been reported. While cholecystectomy is the mainstay treatment for AAC, this might not be the case for HAV induced AAC. For instance, unless there is necrotic gallbladder or persistence of symptoms, the AAC can be managed conservatively in this case. Even though our diagnosis was cleared post-operatively, had we know the diagnosis of HAV induced AAC before, we would still opt for surgery due to the severity and persistence of pain.

Conclusion: More cases should be reported and more studies should be done to further define the presentation and management of HAV induced AAC.

ELIGIBILITY:
Inclusion Criteria:

* acalculous cholecystitis

Exclusion Criteria:

* calculous cholecystitis

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients presenting with symptoms of acute acalculous cholecystitis
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Hepatitis A induced acute acalculous cholecystitis | 1 month
  Laparoscopic cholecystectomy for hepatitis A induced acute acalculous cholecystitis

CONTACTS AND LOCATIONS:
Locations (1):
- University Of balamand, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Publishing a case report